CLINICAL TRIAL: NCT04643236
Title: Increased Knowledge About The Pathogenesis Of Periodontal Disease Improve Oral Hygiene In Patients With Gingivitis-A Blinded Randomised Controlled Clinical Study
Brief Title: Increased Knowledge Improve Oral Hygiene In Patients With Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sadiye Gunpinar, Asst.Prof., Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017/151
Record Dates: First submitted 2020-11-13; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Gingivitis
Keywords: motivational interview; periodontal disease; oral hygiene
MeSH Terms: conditions — Gingivitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: A Single-Centre, Randomised, Parallel Design Controlled Clinical Study
Who Masked: Investigator, Outcomes Assessor
Masking Description: A total of 50 sealed envelopes were prepared in which the group names were written. Following, they were separated in two plastic boxes equally. The group of each participant was recorded by the first author whom the educational intervention was performed (SG). The examiner who performed the clinical process (BM) was unaware of the groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periodontal health educational group (test) (Experimental): 25 subjects diagnosed with gingivitis received periodontal health education session
  Interventions: Behavioral: Periodontal health education session
- oral hygiene motivation group (control) (Active Comparator): 25 subjects diagnosed with gingivitis received standard oral hygiene motivation session
  Interventions: Behavioral: Oral hygiene motivation session

INTERVENTIONS:
Behavioral: Periodontal health education session — This session comprised of a condensed version of motivational interviewing and a periodontal education view/point. First, patients were analysed in terms of expectations from periodontal treatment/oral hygiene practice, knowledge about periodontal diseases and its consequences, daily oral hygiene routine, awareness of the current periodontal status and the main reasons for not doing proper brushing and interproximal cleaning. The same researcher who did not included in the clinic process informed the patients about how periodontal diseases develops, its aetiology, symptoms, consequences and the relationship with the important systemic disorders verbally and via brochure as well. The importance of the patients' own efforts about daily cleaning of the mouth were emphasized. Finally oral hygiene instructions, including brushing and flossing, were demonstrated to each patient after nonsurgical periodontal treatment.
  Arms: periodontal health educational group (test)
Behavioral: Oral hygiene motivation session — Standard oral hygiene instructions, including brushing and flossing, were demonstrated to each patient after nonsurgical periodontal treatment.
  Arms: oral hygiene motivation group (control)

SUMMARY:
Proper plaque control is essential for to maintain oral and general health therefore, improving patient motivation is crucial for to prevent oral diseases including periodontal diseases. The aim of this clinical trial is to evaluate the effect of periodontal health education session (PHES) including the pathogenesis and consequences of periodontal diseases on oral hygiene motivation in patients with gingivitis.

DETAILED DESCRIPTION:
A randomized controlled clinical trial design with 50 subjects (26 Females and 24 males) was carried out in a group of gingivitis patients who underwent periodontal treatment. Subjects were randomly allocated into PHES group (test, n = 25) and standard oral hygiene education group (OHE) (control, n=25). Test group received information about the pathogenesis of periodontal diseases, its consequences, its interaction with systemic diseases and the importance of daily proper cleaning by experienced periodontologist via brochure. Control group received only standard oral hygiene instructions. The Rustogi Modified Navy Plaque index (RMNPI) and papillary bleeding index (PBI) were utilized to evaluate the oral hygiene at baseline and repeated at 1, 3 and 6 months follow-up.

The clinical outcome variables of RMNPI (primary outcome) and PBI (secondary outcome) scores were analysed with Mann Whitney U test. Friedman-Wilcoxon sign ranked test was used for within group comparison. All data were analysed using the Statistical software (SPSS, version 19.0, Chicago, IL, USA). A p-value of <0.05 was accepted as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with gingivitis (no clinical attachment loss) and no previous periodontal treatment,
* non-smokers,
* aged>22 years old and who have a university degree,
* had a visible plaque level > 50%.

Exclusion Criteria:

* Patients having systemic conditions that could affect the healing process and prevent the application of oral hygiene instructions,
* Patients rehabilitated with teeth/implant supported prostheses,
* Patients diagnosed with periodontitis,
* Patients having defective restorations/active teeth related infection or ongoing orthodontic treatment
* Patients who had to be out of the city in a long time during the study period.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Rustogi Modified Navy Plaque index (RMNPI) scores | Measured at Baseline and at 1st-, at 3rd- and at 6th month after nonsurgical periodontal treatment.
  The facial/lingual surfaces of each teeth was divided in nine region and scored as 0: absence of plaque and 1: existence of plaque. The averages of the sum of those scores were evaluated per patient as total (A+B+C+D), gingival margin associated (A+B+C) and interproximal region associated plaque above the margin (D+F). Furthermore, the indicator of proper interproximal cleaning surface area (A+C+D+F) was also evaluated per patient.
  The change in RMNPI scores between all time intervals were evaluated and compared between study groups.

SECONDARY OUTCOMES:
Change in Papillary bleeding index (PBI) scores | Measured at Baseline and at 1st-, at 3rd- and at 6th month after nonsurgical periodontal treatment.
  Each papilla region was scored and the mean of those scores were recorded as PBI per patient. Accordingly, 0: no bleeding; 1: a single isolated bleeding point; 2: several isolated bleeding points; 3: interdental triangle fills with blood soon after probing; 4: intense bleeding occurs immediately after probing through the gingival margin.
  The change in PBI scores between all time intervals were evaluated and compared between the study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University, Faculty of Dentistry, Department of Periodontology, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available now.